CLINICAL TRIAL: NCT03720639
Title: Confirm Rx™ Versus Reveal LINQ™ -Which is More Reliable in Data Transmission? A Randomized Clinical Study
Brief Title: Confirm Rx™ Versus Reveal LINQ™ - Which is More Reliable in Data Transmission? A Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sparrow Clinical Research Institute (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, John H. Ip, M.D., Medical Director, Sparrow Clinical Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 41618
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Arrythmias; Syncope; Atrial Fibrillation; Atrial Flutter; Tachycardia; Stroke
Keywords: Implantable Loop Recorder; Implantable Cardiac Monitor; Cryptogenic Stroke
MeSH Terms: conditions — Syncope; Atrial Fibrillation; Atrial Flutter; Tachycardia; Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Abbott, Inc Confirm Rx™ (Active Comparator): Every other consenting subject will receive the Abbott Inc. Confirm Rx™ device.
  Interventions: Device: Abbott, Inc Confirm Rx™ versus Medtronic, Inc Reveal LINQTM
- Medtronic, Inc Reveal LINQTM (Active Comparator): Every other consenting subject will receive the Medtronic, Inc. Reveal LINQTM.
  Interventions: Device: Abbott, Inc Confirm Rx™ versus Medtronic, Inc Reveal LINQTM

INTERVENTIONS:
Device: Abbott, Inc Confirm Rx™ versus Medtronic, Inc Reveal LINQTM — Comparing reliability and timeliness in data transmission between two implantable cardiac monitors.

SUMMARY:
This study will compare the reliability and timeliness in data transmission of the Abbott Confirm Rx™ loop recorder with the Medtronic Reveal LINQ™ loop recorder.

DETAILED DESCRIPTION:
Implantable cardiac monitor (ICM) is an invaluable tool for diagnosing cardiac arrhythmia (1). Cryptogenic stroke, unexplained syncope and arrhythmia diagnosis are the most common indication for long term cardiac monitoring device. (2, 3). Reveal LINQTM (Medtronic, Inc.) is widely used for all of these purposes in the country. We have previously reported the use of Reveal XT in the use of atrial fibrillation (AF) surveillance in patient's post-AF ablation (2). We indicated that ICM is useful in long term monitoring of atrial arrhythmia in patients at risk of atrial fibrillation. Crystal AF (4) study also showed the importance of using ICM in detecting occult AF in patients with cryptogenic stroke in a timely manner so that appropriate treatment can be prescribed. The key to the success of ICM rest on how timely and reliable the ICM data can be transmitted to physician's office immediately after an arrhythmic events so the data can be analyzed and treatment rendered. Reveal LINQTM data transmission consists of two steps: 1. Data needs to be download into the MyCareLink™ monitor (scheduled daily at 2 am in the morning and monitor needs to be in the within 6 feet proximity of the patient) 2. MyCareLink™ monitor to be connected to the 3 G cellular network for the data transmission. (Fig 1). In cases of patient activated events, data transmission utilizes similar pathway.

We have reported significant delay in data transmission in the Reveal LINQTM occurs frequently and failure to connect among the Reveal LINQTM, MyCareLink™ monitor and the cellular network is the main reason for data transmission disruption and critical data could be concealed for an extended periods. To illustrate the importance of timely transmission of patient data, a Reveal LINQTM was implanted in a 54-year-old gentle man with past medical history of recurrent syncope. On 8/12/2017 the patient developed new onset dizziness and 6 seconds sinus pause was recorded by the device. However, a connection problem of MyCarelinkTM system made data unavailable until next scheduled office visit on 11/15/2017. The physician was notified on the same day and a pacemaker was implanted on the following day, almost 3 months after his significant arrhythmic events.

The newer generation of ICM such as Confirm Rx™ (Abbott, Inc) is connected directly to a patient's existing smartphone using the Bluetooth technology. By allowing patients to record and transmit symptoms with the mobile app, Confirm Rx™ ICM brings continuous remote monitoring to patients without the need for a home-based monitor (Fig 2). It is unclear which technologies offers faster and more reliable transmission of critical patient information to physician office so timely treatment can be provided. We therefore propose a pilot randomized study comparing Confirm Rx™ and Reveal LINQTM in the reliability and timeliness in data transmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient is willing and able to provide written informed consent
* Patient is willing and able to comply with the protocol, including follow-up visits and MyCareLink™ and Merlin™ transmissions (standard of care)
* Candidates for implantable cardiac monitor

Exclusion Criteria:

* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a study manager
* Patient has existing IPG, ICD, CRT-D or CRT-P device
* Adequate sensing in one week post implant. If sensing not adequate, patient will be in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Time from arrhythmic events to time of physician notification | 12 months
Time from activated events to time of physician notification | 12 months

SECONDARY OUTCOMES:
Time from arrhythmic events to time of intervention if any | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John H Ip, MD, Principal Investigator — Sparrow Hospital
Locations (2):
- United States (2):
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Munson Medical Center, Traverse City, Michigan

IPD SHARING:
Plan to Share IPD: No